CLINICAL TRIAL: NCT03733067
Title: Phase 1/2 Randomized, Double-Blind, Placebo-Controlled Study of Safety and Efficacy of Abatacept for Treating Chronic Cytopenia in Cytotoxic T-lymphocyte Antigen 4 (CTLA4) Haploinsufficiency
Brief Title: Safety and Efficacy of Abatacept for Treating Chronic Cytopenia in Cytotoxic T-Lymphocyte Antigen 4 (CTLA4) Haploinsufficiency
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: No enrollment
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 190015; 19-I-0015
Record Dates: First submitted 2018-11-06; First posted 2018-11-07 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: CTLA4 Haploinsufficency; Chronic Cytopenia
Keywords: Regulatory T Cells; T-cell hyperactivation; Autoimmune Cytopenia; Adult Rheumatoid Arthritis; Juvenile Idiopathic Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis, Juvenile | interventions — Abatacept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- abatacept (Experimental): Adult and pediatric dosing will be based on weight per protocol
  Interventions: Drug: abatacept
- placebo (Placebo Comparator): will be given as the same IV volume as abatacept
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: abatacept — Double-blind, placebo-controlled, intra-patient dose-escalation trial of abatacept for treating cytopenia in CTLA4 deficiency. Abatacept or placebo will be administered for 3 doses over 30 days, followed by 5 more months of administration at double the initial dose. If the participant s hematologic parameters normalize at Day 120 or onwards, the investigator may taper or discontinue concomitant medications aimed at treating cytopenia.
  Arms: abatacept
Other: Placebo — Saline packaged identically to abatacept, with volume matching that of the abatacept dosing by weight, and will be administered via IV infusion identically to abatacept
  Arms: placebo

SUMMARY:
Background:

CTLA4 stands for cytotoxic T-lymphocyte antigen-4. It is a protein the body makes naturally to check its immune system from attacking itself. Some people don t produce enough CTLA4 protein, causing problems due to overactive immune system such as big spleens, repeated lung infections, breathing problems, stomach and intestine symptoms as well as inflamed brain and nerve problems. Many have problems with their bone marrow causing low numbers of blood cells like platelets, red blood cells or white blood cells, which is called cytopenia. Researchers want to see if the drug abatacept can treat cytopenias by replacing the missing protein CTLA4.

Objective:

To see if abatacept is safe and helps treat cytopenias caused by CTLA4 deficiency.

Eligibility:

People ages 8-65 years who have CTLA4 deficiency with cytopenia

Design:

Participants will be screened with medical history, medication review, physical exam and blood and urine tests. They will continue their current medications and may start taking antibiotics daily. Participants will receive either abatacept or placebo through a vein for 6 months. The study team will not know if you are receiving the study drug or the placebo

Women who can become pregnant must agree to use birth control measures.

Men who get someone pregnant during the study will be asked to collect information and have the partner contact the study team.

Participants will undergo the following procedures before starting the study and at the completion:

* radiology scans of body and brain
* heart and lung function tests
* Bone marrow examination by a needle inserted into the hip bone to remove a small amount of tissue to study.
* Participants may have a small camera on a long, thin tool passed down the throat into the stomach and small intestine for evaluation of their gut.
* Questionnaires about their disease, symptoms and quality of life

Over 6 months, participants will have regular study visits and get 8 doses of the study drug or a placebo by intravenous injection. They will repeat some of the same tests done earlier at the end of the study at assess response.

About 1 month after the last study drug visit, participants will have a final study visit.

Some participants may join a treatment extension for the study drug abatacept with no placebo. They will sign a separate consent form for this.

DETAILED DESCRIPTION:
Rare heterozygous mutations in cytotoxic T-lymphocyte antigen-4 (CTLA4) lead to a monogenetic defect that presents with a heterogeneous clinical phenotype of recurrent infections, lymphoproliferation, autoimmunity, and lymphocytic infiltration of target organs. Management is challenging and focuses on treating infections, autoimmune complications, and end organ damage due to lymphocytic infiltrates. Experience with the natural history of the disease and therapies for underlying complications are limited. There is no established standard of care for these patients.

Abatacept is a biologically engineered CTLA4-mimetic that is approved as an intravenous (IV) infusion to treat adult rheumatoid arthritis, adult psoriatic arthritis, and juvenile idiopathic arthritis. Given that abatacept mimics CTLA4 function, we hypothesize that the drug will prevent T-cell hyper-activation, restore regulatory T-cell function, and thereby treat the autoimmune and immune dysregulatory manifestations of CTLA4 deficiency.

This study is a phase 1/2, double-blind, randomized, intra-patient dose-escalation, placebo-controlled trial designed to evaluate the safety and efficacy of abatacept in participants with CTLA4 deficiency and cytopenia. Participants will come to the NIH Clinical Center monthly for 210 days to receive infusions of study agent or placebo and to undergo safety and research evaluations, including blood draw for cytopenia evaluation and scoring of disease severity. Before and after the treatment period, participants will also have imaging, pulmonary function testing, bone marrow biopsy, and endoscopy (symptomatic participants only). Primary endpoints will be evaluated at Day 210. After completing the blinded treatment trial, participants will be offered the option to enroll in a 6-month open-label extension study for long-term safety evaluation of abatacept.

ELIGIBILITY:
* INCLUSION CRITERIA:

Individuals must meet all of the following criteria to be eligible for study participation:

1. Age 8-65 years.
2. Documented CTLA4 mutation (requires documentation of confirmed mutation via Sanger sequencing at a laboratory approved by the Clinical Laboratory Improvement Amendments [CLIA]).
3. At least one of the following established hematologic abnormalities during the past 6 months (including results from outside CLIA-certified laboratories) prior to screening:

   * ANC < 750 cells/microL.
   * Platelet count < 75,000 cells/microL.
   * Hemoglobin < 7.5 g/dL.
4. The above mentioned hematologic abnormalities should require active treatment with steroids, immunomodulatory agents (e.g., mycophenolate mofetil, cyclosporine, tacrolimus, mercaptopurine, methotrexate, sirolimus, high dose intravenous immunoglobulin [IVIG]), and/or other agents (e.g., TPO agonists) for at least 60 days prior to screening.
5. The dose of any concomitant medication(s) aimed at treating cytopenia should be stable in the 60 days prior to screening. Stable is defined as:

   * No new concomitant medications for cytopenia were initiated.
   * No dose increase of the medication was required.
6. Did not receive blood product transfusions within 30 days prior to screening.
7. Did not receive abatacept within 60 days prior to screening.
8. Did not receive rituximab within 3060 days of screening.
9. Did not receive alemtuzumab at any time.
10. Has access to healthcare provider at home.
11. Able to provide informed consent.
12. Willing to allow storage of biological specimens for future use in medical research.
13. Females of childbearing potential must agree to use appropriate birth control methods when engaging in sexual activities that can result in pregnancy, beginning Day -30 through 30 days after the last dose of study agent. Appropriate methods should include 2 forms of contraception, one from each of the following categories:

    * Hormonal contraception or placement of an intrauterine device or intrauterine system.
    * Barrier method: Condom or occlusive cap (diaphragm or cervical/vault cap) with a spermicide.

EXCLUSION CRITERIA:

Patients meeting any of the following criteria are not eligible for this study:

1. History of hypersensitivity to abatacept.
2. Any live vaccines (including attenuated live vaccines) within 6 weeks of screening.
3. History of acquired immunodeficiency diseases, including a positive HIV polymerase chain reaction (PCR) test result.
4. Untreated chronic hepatitis B (positive PCR) or hepatitis C (positive PCR) infection. Patients with chronic hepatitis must be on medical treatment for at least 3 months before screening and have evidence of decreased viral loads after starting treatment.
5. EBV viral load > 4log on 2 or more laboratory checks greater than 1 month apart and within 6 months of screening.
6. History of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past 5 years, regardless of evidence of local recurrence or metastases.
7. Current active infectious disease (bacterial or fungal) including evidence of tuberculosis (TB) infection as defined by a positive QuantiFERON TB-Gold test. Test results within the past 6 months will be accepted. If presence of latent TB is established, then treatment must be completed before the patient can be considered for enrollment. The patient may also be considered for enrollment after completing treatment of any other active bacterial or fungal infection.
8. Contraindication to PFT or CT scan.
9. Pregnancy or breastfeeding.
10. Any condition that, in the opinion of the investigator, contraindicates participation in this study.

Ages: 8 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-11-30 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
assess safety and tolerability of abacept given at double doses | To be measured at day 210
  All safety parameters (including possibly to definitely related AEs and SAEs, physical exam, vital signs, ECG, safety laboratories [hematology, blood chemistry, urinalysis]) and incidence and severity of infections at initial and doubled doses of abatacept at Day 210.
Clinical Efficacy of abatacept in normalizing cytopenias | To be measured at day 210
  A complete response defined by the normalization of all listed hematologic parameters:A) ANC > 1,000 cells/microliter; andB) Platelet count > 100,000 cells/microliter; andC) Hemoglobin > 10 g/dLParameters will be measured at Day 210 and must be met without any transfusions and concomitant medications (immunomodulatory therapy, exogenous growth factor, steroids, hematopoietic/TPO mimetic agent) aimed at treating cytopenias during the past 28 days.

SECONDARY OUTCOMES:
measure of time to cytopenia recurrence | From initiating the taper or discontinuation of concomitant medications while on treatment
Clinical efficacy of abatacept in improving but not normalizing cytopenais | To be measured at Day 210
  Partial hematologic response defined as an improvement in one or more of the listed parameters but not meeting complete hematologic response:A) ANC: a 100% increase from baseline or an ANC >= 750 cells/microL.B) Platelet: for baseline count >= 20,000/microL but < 75,000/microL: a 100% increase in platelet count or a platelet count > 75,000/ (Micro)L; for baseline platelet count < 20,000/micro: a 100% increase in platelet count or a platelet count > 20,000/microL.C) Any increase in hemoglobin by 2 g/dL.All of the parameters will be measured at Day 210 and must be met without any transfusions and concomitant medications (immunomodulatory therapy, exogenous growth factor, steroids, hematopoietic/TPO mimetic agent) aimed at treating cytopenias during the past 28 days. OR A normalization of hematologic parameters as defined in the primary endpoint AND a dose reduction or discontinuation of baseline concomitant medications.

CONTACTS AND LOCATIONS:
Overall Officials: Gulbu Uzel, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lo B, Zhang K, Lu W, Zheng L, Zhang Q, Kanellopoulou C, Zhang Y, Liu Z, Fritz JM, Marsh R, Husami A, Kissell D, Nortman S, Chaturvedi V, Haines H, Young LR, Mo J, Filipovich AH, Bleesing JJ, Mustillo P, Stephens M, Rueda CM, Chougnet CA, Hoebe K, McElwee J, Hughes JD, Karakoc-Aydiner E, Matthews HF, Price S, Su HC, Rao VK, Lenardo MJ, Jordan MB. AUTOIMMUNE DISEASE. Patients with LRBA deficiency show CTLA4 loss and immune dysregulation responsive to abatacept therapy. Science. 2015 Jul 24;349(6246):436-40. doi: 10.1126/science.aaa1663. PMID 26206937
- [Background] Lee S, Moon JS, Lee CR, Kim HE, Baek SM, Hwang S, Kang GH, Seo JK, Shin CH, Kang HJ, Ko JS, Park SG, Choi M. Abatacept alleviates severe autoimmune symptoms in a patient carrying a de novo variant in CTLA-4. J Allergy Clin Immunol. 2016 Jan;137(1):327-330. doi: 10.1016/j.jaci.2015.08.036. Epub 2015 Oct 21. No abstract available. PMID 26478010
- [Background] Salman J, Ius F, Knoefel AK, Sommer W, Siemeni T, Kuehn C, Tudorache I, Avsar M, Nakagiri T, Preissler G, Hatz R, Greer M, Welte T, Haverich A, Warnecke G. Association of Higher CD4+ CD25high CD127low , FoxP3+ , and IL-2+ T Cell Frequencies Early After Lung Transplantation With Less Chronic Lung Allograft Dysfunction at Two Years. Am J Transplant. 2017 Jun;17(6):1637-1648. doi: 10.1111/ajt.14148. Epub 2017 Jan 24. PMID 27931084
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2019-I-0015.html